CLINICAL TRIAL: NCT03951883
Title: Does Increased Egg Consumption Have Cognitive and Neural Benefits in Food Insecure, At-risk Adolescents?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Principal Investigator, Martin Binks, Associate Professor, Texas Tech University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TTUIRB2019-160
Record Dates: First submitted 2019-05-10; First posted 2019-05-16 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Adolescents With Food Insecurity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Typical Diet (TD) (Active Comparator): Participants will be instructed to continue habitual dietary intake.
  Interventions: Other: Typical diet
- Increased Egg Consumption (IE) (Experimental): Participants will be prescribed an additional 2 eggs per day to their diet.
  Interventions: Other: Increased Egg Consumption

INTERVENTIONS:
Other: Increased Egg Consumption — Subjects will be instructed to use a weekly food purchase supplement for inclusion of 2 additional eggs per day to be added to subject's typical daily diet.
  Arms: Increased Egg Consumption (IE)
Other: Typical diet — Subjects will be instructed to maintain their current dietary patterns.
  Arms: Typical Diet (TD)

SUMMARY:
Quality nutrient intake is essential for proper development and well-being of children in all aspects of health, including cognitive development. Eggs are of particular interest based on potential cognitive and neurological benefits due in part to significant concentrations of choline and lutein. While overall, choline and lutein have received considerable attention in the literature in relation to cognition and brain function, most studies involving intake in young adults have had short intervention periods ranging from 90 minutes to 3 days. Food insecurity has been associated with decreased academic performance. Given that populations with food insecurity have limited resources to direct towards nutrition, identifying how a widely available, highly versatile and largely affordable source of nutrients (i.e. eggs) may have favorable impacts on cognitive function and brain function will be valuable in informing public health recommendations in this at-risk population. As such the investigators will examine whether an increased egg consumption dietary prescription can have positive effects on functional activity (i.e. fMRI) during an Eriksen-Flanker task, anatomical changes in the brain (i.e. DTI, MRI), and cognitive abilities as measured by the Stop Signal Reaction Time task, Operation Span task, Raven's Progressive Matrices and the Boston Naming Task.

ELIGIBILITY:
Inclusion Criteria:

* Age: 13-19 years.
* Household has food security status of low or very low as designated by scoring 2-6 raw score using the U.S. Household Food Security Survey Module: Six-Item Short Form.

Exclusion Criteria:

* Participants unable or unwilling to provide informed consent.
* Participants with motor, visual or hearing impairment.
* Participants with current severe psychiatric illnesses (e.g. psychosis, schizophrenia, bipolar disorders, depression)
* Participants with history of psychiatric hospitalization.
* Participants with habitual egg consumption (past 3 months) of 4 eggs per week or more
* Unable or unwilling to consume required study meals for any reason (e.g. dietary restrictions, allergies, or aversions to any of the food items used in the study).
* History of liver or kidney disease, cardiovascular disease, hematologic disease, metabolic disease, Epilepsy (or other seizure disorder) or malignant tumor
* Currently taking (or have taken in the past 4 weeks) any anti-anxiolytic, anti-epileptic, or anti-depression medications
* Currently taking (or have taken in the past 4 weeks) any proton pump inhibitor medications
* History of any cognitive disorder, medical and/or psychological conditions and/or medications affecting cognition
* Participants with contraindications for MRI scanning.

  1. aneurism clips
  2. any implanted medical devices (pacemaker, neurostimulator)
  3. known pregnancy
  4. shrapnel in body or any injury to eye involving metal
  5. any ferrous metal in body

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Comparison of functional activity during Eriksen-Flanker Task | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Changes in regional brain activation during an fMRI scan.
Comparison of grey matter anatomical change | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Grey density as measured by MRI
Comparison of white matter connectivity change | Baseline (pre-intervention) and 12 weeks (post-intervention)
  White matter connectivity as measured by diffusion tensor imaging
Comparison of cognitive battery performance change | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Cognitive performance as measured by stop signal reaction time task
Comparison of cognitive battery performance change | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Cognitive performance as measured by operation span task
Comparison of cognitive battery performance change | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Cognitive performance as measured by Raven's Progressive Matrices
Comparison of cognitive battery performance change | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Cognitive performance as measured by Boston Naming Task
Comparison of Eriksen-Flanker Task performance change | Baseline (pre-intervention) and 12 weeks (post-intervention)
  Eriksen-Flanker task performance compared using the drift diffusion model

CONTACTS AND LOCATIONS:
Overall Officials: Martin Binks, PhD, Principal Investigator — Texas Tech University- Department of Nutritional Sciences
Locations (2):
- United States (2):
  - Texas Tech Neuroimaging Institute, Lubbock, Texas
  - Nutrition & Metabolic Health Initiative, Lubbock, Texas